CLINICAL TRIAL: NCT00215605
Title: A Phase 1 Dose-Escalation Study of the Safety and Pharmacokinetics of XL184 Administered Orally to Subjects With Advanced Malignancies
Brief Title: Study of XL184 (Cabozantinib) in Adults With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL184-001; NCT00354289 (obsolete NCT alias)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Lymphoma; Cancer; Thyroid Carcinoma
Keywords: Advanced Malignancies; Solid Tumor; Medullary Thyroid Cancer
MeSH Terms: conditions — Lymphoma; Neoplasms; Thyroid Neoplasms; Carcinoma, Medullary

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: XL184

INTERVENTIONS:
Drug: XL184 — Flavored liquid suspension or gelatin capsules supplied in 25-mg and 100-mg strengths; daily dosing or intermittent schedule (daily dosing followed by dosing holiday in cycles)

SUMMARY:
The purpose of this study is to determine the best and safest dose of XL184 administered orally. XL184 is a new chemical entity that inhibits VEGFR2, MET and RET, kinases implicated in tumor formation, growth and migration. To determine the highest safe dose, subjects will receive different amounts of the drug. The first group of subjects will receive the lowest dose of XL184. As long as no medically unacceptable side effects are noted, the dose will be increased for the next group. When the maximum tolerated dose (MTD) is reached, at least 20 subjects with Medullary Thyroid Cancer (MTC) will be enrolled to evaluate the effect of XL184 in this population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced malignancy (solid tumor or lymphoma) that is metastatic or unresectable for which standard curative measures do not exist or are no longer effective
* Eastern Cooperative Oncology Group (ECOG) performance status </= 2
* Life expectancy greater than 3 months
* Adequate organ and marrow function
* Written informed consent
* Use of acceptable methods of contraception during the course of the study and for 3 months after completion of study
* In the MTD expanded cohort: at least 20 subjects with metastatic and/or advanced/locally recurrent Medullary Thyroid Cancer not appropriate for surgical resection with measurable disease as defined by RECIST

Exclusion Criteria:

* Chemotherapy, immunotherapy or radiation within 4 weeks (or nitrosoureas or mitomycin C within 6 weeks) before the first scheduled dose of XL184
* Administration of an investigational drug within 30 days of the first dose of XL184
* Subject has not recovered from adverse events due to investigational agents or other medications administered more than 4 weeks before study enrollment
* Known brain metastases
* Uncontrolled intercurrent illness
* Pregnancy or breastfeeding
* Known HIV positive
* Known allergy or hypersensitivity to any of the components of the XL184 formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2005-09; Primary Completion 2011-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, maximum tolerated dose (MTD), and dose-limiting toxicity of oral administration of XL184 | Assessed during periodic visits
Evaluate plasma pharmacokinetics and estimate renal elimination of oral administration of XL184 | Assessed during periodic visits

SECONDARY OUTCOMES:
Long-term safety/tolerability of XL184 after oral administration for up to 1 year | Assessed during periodic visits
Evaluate preliminary tumor response after repeated XL184 administration | Assessed during periodic visits
In MTD expanded cohort: Progression-free survival and duration of response in subjects with advanced or recurrent medullary thyroid cancer | Assessed during periodic visits

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Univ. of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Kurzrock R, Atkins J, Wheler J, Fu S, Naing A, Busaidy N, Hong D, Sherman S. Tumor marker and measurement fluctuations may not reflect treatment efficacy in patients with medullary thyroid carcinoma on long-term RET inhibitor therapy. Ann Oncol. 2013 Sep;24(9):2256-61. doi: 10.1093/annonc/mdt177. Epub 2013 May 14. PMID 23676418
- [Derived] Kim KB, Cabanillas ME, Lazar AJ, Williams MD, Sanders DL, Ilagan JL, Nolop K, Lee RJ, Sherman SI. Clinical responses to vemurafenib in patients with metastatic papillary thyroid cancer harboring BRAF(V600E) mutation. Thyroid. 2013 Oct;23(10):1277-83. doi: 10.1089/thy.2013.0057. Epub 2013 Jul 17. PMID 23489023
- [Derived] Kurzrock R, Sherman SI, Ball DW, Forastiere AA, Cohen RB, Mehra R, Pfister DG, Cohen EE, Janisch L, Nauling F, Hong DS, Ng CS, Ye L, Gagel RF, Frye J, Muller T, Ratain MJ, Salgia R. Activity of XL184 (Cabozantinib), an oral tyrosine kinase inhibitor, in patients with medullary thyroid cancer. J Clin Oncol. 2011 Jul 1;29(19):2660-6. doi: 10.1200/JCO.2010.32.4145. Epub 2011 May 23. PMID 21606412